CLINICAL TRIAL: NCT02720484
Title: Phase II Study of Nivolumab (Anti-PD-1 Antibody) for Treatment of Metastatic Adrenocortical Carcinoma
Brief Title: Nivolumab in Treating Patients With Metastatic Adrenocortical Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study did not meet first stage requirements of interim analysis
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 15E01; STU00202153 (CTRP (Clinical Trial Reporting Program)); NU 15E01 (Other: Northwestern University); P30CA060553 (NIH); NCI-2016-00194 (Other: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2016-03-16; First posted 2016-03-28 (Estimated); Results first posted 2019-05-01 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-02

CONDITIONS: Metastatic Carcinoma in the Adrenal Cortex; Recurrent Adrenal Cortex Carcinoma; Stage III Adrenal Cortex Carcinoma; Stage IV Adrenal Cortex Carcinoma
MeSH Terms: conditions — Adrenal Cortex Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Nivolumab) (Experimental): Patients receive nivolumab IV over 30 minutes every 2 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Nivolumab

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; ONO-4538; Opdivo

SUMMARY:
The primary objective will be to assess overall response rate of nivolumab in patients with metastatic or locally advanced adrenocortical carcinoma. Nivolumab was recently approved by U.S. Food and Drug Administration (FDA) for the treatment of advanced melanoma, non-small cell lung cancer and renal cell carcinoma. It is considered investigational for the treatment of advanced or refractory adrenocortical carcinoma. "Investigational" means that the drug is not approved by the USFDA or not approved for the indication under investigation. Nivolumab could shrink adrenocortical carcinoma but it could also cause side effects. Researchers hope to learn if the study drug will shrink the cancer and hopefully to relieve symptoms that are related to the cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess overall response rate of nivolumab in patients with metastatic or locally advanced adrenocortical carcinoma (ACC).

SECONDARY OBJECTIVES:

I. To assess the progression free survival defined as time from date of first nivolumab infusion until date of death or evidence of progression of disease as assessed by computed tomography (CT) imaging every 8 weeks according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria 1.1.

II. To assess the overall survival defined as time from date of first nivolumab infusion until death of patients with metastatic or locally advanced ACC.

III. To assess the safety and tolerability profile of nivolumab described by number, frequency, and severity of adverse events according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.3 assessed every 2 weeks while patients are on therapy.

TERTIARY OBJECTIVES:

I. To assess the overall response rate, progression free survival and overall survival according to tumor programmed cell death 1 ligand 1 (PD-L1) and programmed cell death 1 ligand 2 (PD-L2) expression.

II. To assess the overall response rate, progression free survival and overall survival according to serum interleukin levels and peripheral T cell profile levels.

III. To measure humoral and cellular responses to tumor antigens on serum samples by measuring the levels of cytokines (ie, interleukin [IL] -2, IL-6, IL-8, IL-10, IL-18, interferon [IFN] gamma and tumor necrosis factor [TNF]-alpha) and peripheral blood lymphocyte phenotype.

OUTLINE:

Patients receive nivolumab intravenously (IV) over 30 minutes every 2 weeks in the absence of disease progression or unacceptable toxicity, or withdrawal of consent.

After completion of study treatment, patients are followed up every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed stage IV or unresectable locally advanced adrenocortical carcinoma
* Patients must have disease progressing after treatment with at least one line of therapy including mitotane and/or chemotherapy; Note: patients declining first line treatment with mitotane and/or chemotherapy based on limited efficacy are also eligible for this study
* Patients must have measurable disease according to the standard RECIST version 1.1; CT scans or magnetic resonance imaging (MRIs) used to assess the measurable disease must have been completed within 28 days prior to registration
* Patients must exhibit an Eastern Cooperative Oncology Group (ECOG) performance status of 0-3
* Leukocytes >= 2,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Hemoglobin >= 9 g/dL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 × institutional upper limit of normal (ULN) (except patients with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
* Aspartate transaminase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine transferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN
* Serum creatinine of < 3.0 x ULN (upper limit of normal) or creatinine clearance (CrCl) > 30 mL/minute (using Cockcroft/Gault formula below)
* Patients with history of central nervous system (CNS) metastases are eligible if CNS disease has been radiographically and neurologically stable for at least 6 weeks prior to study registrations and do not require corticosteroids (of any dose) for symptomatic management
* Females of childbearing potential (FOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 72 hours prior to the start of study drug; NOTE: a FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria: has not undergone a hysterectomy or bilateral oophorectomy; has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)
* FOCBP must agree to follow instructions for method(s) of contraception (e.g. hormonal or barrier method of birth control; abstinence) for the duration of treatment with nivolumab plus 5 half-lives of nivolumab (19 weeks) plus 30 days (duration of ovulatory cycle) for a total of 23 weeks post-treatment completion
* Males who are sexually active with women of childbearing potential (WOCBP) must agree to follow instructions for method(s) of contraception (e.g. hormonal or barrier method of birth control; abstinence) for the duration of treatment with nivolumab plus 5 halflives of the study drug (19 weeks) plus 90 days (duration of sperm turnover) for a total of 31 weeks days post-treatment completion
* Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study are not eligible
* Patients who have not recovered to =< grade 1 from adverse events due to agents administered more than 4 weeks earlier are not eligible
* Patients may not be receiving any other investigational agents
* Patients who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to nivolumab are not eligible
* Patients should be excluded if they have had prior treatment with an anti-PD1 or anti-PD-L1. Please contact principal investigator, Benedito Carneiro, for specific questions on potential interactions
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including chronic prolonged systemic corticosteroids (defined as corticosteroid use of duration one month or greater), should be excluded; these include but are not limited to patients with a history of:

  * Immune related neurologic disease
  * Multiple sclerosis
  * Autoimmune (demyelinating) neuropathy
  * Guillain-Barre syndrome
  * Myasthenia gravis
  * Systemic autoimmune disease such as systemic lupus erythematosus (SLE)
  * Connective tissue diseases
  * Scleroderma
  * Inflammatory bowel disease (IBD)
  * Crohn's
  * Ulcerative colitis
  * Patients with a history of toxic epidermal necrolysis (TEN)
  * Stevens-Johnson syndrome
  * Anti-phospholipid syndrome; Note: subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* Any condition requiring systemic treatment with corticosteroids (> 10mg daily prednisone equivalents) or other immunosuppressive medications within 14 days prior to first dose of study drug; Note: inhaled steroids and adrenal replacement steroid doses > 10mg daily prednisone equivalents are permitted in the absence of active autoimmune disease; a brief (less than 3 weeks) course of corticosteroids for prophylaxis (eg, contrast dye allergy) or for treatment of non-autoimmune conditions (eg, delayed-type hypersensitivity reaction caused by a contact allergen) is permitted
* Patients who have an uncontrolled intercurrent illness including, but not limited to any of the following, are not eligible
* Hypertension that is not controlled on medication (Note: hypertension is defined as blood pressure >= 140/90)
* Ongoing or active infection requiring systemic treatment
* Symptomatic congestive heart failure
* Unstable angina pectoris
* Cardiac arrhythmia
* Psychiatric illness/social situations that would limit compliance with study requirements
* Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints
* Female patients who are pregnant or nursing are not eligible
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for at least three years
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS) is not permitted
* Any known positive test for hepatitis B or hepatitis C virus indicating acute or chronic infection is not permitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-03-30 (Actual); Primary Completion 2017-04-17 (Actual); Study Completion 2018-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benedito Carneiro, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio

REFERENCES:
- [Derived] Carneiro BA, Konda B, Costa RB, Costa RLB, Sagar V, Gursel DB, Kirschner LS, Chae YK, Abdulkadir SA, Rademaker A, Mahalingam D, Shah MH, Giles FJ. Nivolumab in Metastatic Adrenocortical Carcinoma: Results of a Phase 2 Trial. J Clin Endocrinol Metab. 2019 Dec 1;104(12):6193-6200. doi: 10.1210/jc.2019-00600. PMID 31276163

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened for accrual on March 22 2016 with an accrual goal of up to 33 patients. The first patient started treatment March 30, 2016. Accrual was suspended on December 5, 2016 after the first 10 patients were enrolled for Interim Analysis. The study was closed permanently on May 24 2017 with no additional patients enrolled.
Period: Treatment on Study
Arm/Group | Treatment (Nivolumab)
Started | 10
Reached 1st Response/2 Cycles | 7
Treated Cycle 3 | 4
Completed | 4
Not Completed | 6
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Progressive Disease | 4
Period: Follow Up for 2 Years
Arm/Group | Treatment (Nivolumab)
Started (2 patients died before entering follow up period and 1 patient withdrew consent.) | 7 (All patients that receive at least one treatment on study go into follow up.)
Completed | 1
Not Completed | 6
Not completed — Withdrawal by Subject | 1
Not completed — Death | 3
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall Response Rate of nivolumab treatment for patients with metastatic adrenocortical carcinoma will be measured per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI scans every 8 weeks:
  Complete Response (CR) = disappearance of all target lesions. Partial Response (PR) >=30% decrease in the sum of the longest diameter of target lesions (should be confirmed 8 weeks after initial response otherwise considered unconfirmed PR).
  Stable Disease, neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study.
  Progressive Disease, defined as having at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions..
Time Frame: From the start of treatment and every 8 weeks/2 cycles with a range of cycles attempted 1-15.
Population: All patients that received one dose of nivolumab were evaluable for this objective.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 10
Participants
  Complete Response | 0
  Unconfirmed Partial Response | 1
  Stable Disease | 2
  Progressive Disease | 6
  NE | 1

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression Free Survival (PFS) of nivolumab treatment in patients with metastatic adrenocortical carcinoma is defined as the duration of time from start of treatment to time of documented progression or death, whichever comes first. It will measured per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI scans every 8 weeks.
Time Frame: From start of treatment and every 8 weeks/2 cycles until progressive disease or death. Median follow up of 4.5 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 10
Months | 1.8 [0.1 to 4.3]

3. Secondary Outcome: Overall Survival (OS) at 3 Months and 6 Months
Description: Overall Survival (OS) of nivolumab treatment in patients with metastatic adrenocortical carcinoma and will be defined as the duration of time from treatment initiation until death. OS will be assessed as the percentage of patients alive at 3 months and at 6 months from initiation of treatment on study.
Time Frame: At 3 months and 6 months from the initiation of treatment
Measure: Number (95% Confidence Interval); unit: percentage of patients alive
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 10
percentage of patients alive
  3 months | 79 [14 to 90]
  6 months | 56 [8 to 88]

4. Secondary Outcome: Toxicity of Nivolumab
Description: Safety and tolerability profile of Nivolumab will be assessed by describing by number, frequency, and severity of Adverse Events (AEs) according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.3. All AEs that were considered related to Nivolumab were collected and are shown below. Patients with multiple events in the same category are counted only once in that category. Patients with events in more than one category are counted in each of those categories. Categories with no events are not shown.
  In general AEs will be graded according to the following:
  Grade 1 = Mild AE Grade 2= Moderate AE Grade 3 = Severe AE Grade 4 = Life-threatening or disabling AE Grade 5 = Death related to AE
Time Frame: From treatment initiation, twice every Cycle (every 14 days) while on treatment, up to 12 weeks after final dose. Range of cycles completed 1-15 (1 Cycle=28 days)
Measure: Number; unit: participants
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 10
participants
  Rash Grade 1-2 | 3
  Nausea Grade 1-2 | 1
  Cough Grade 1-2 | 2
  Fatigue Grade 1-2 | 3
  ALT Increase Grade 1-2 | 1
  ALT Increase Grade 4 | 1
  AST Increase Grade 1-2 | 2
  AST Increase Grade 3 | 1
  Bilirubin Elevation Grade 1-2 | 2
  Hypokalemia Grade 3 | 1
  Dehydration Grade 3 | 1
  Mucositis Grade 1-2 | 3
  Tremor Grade 3 | 1
  Edema Grade 1-2 | 2
  Immune Pneumonitis Grade 3 | 1
  Immune Hepatitis Grade 3 | 1

5. Other Pre Specified Outcome: Levels of Cytokines
Description: Humoral and cellular responses to tumor antigens on serum samples will be evaluated by measuring the levels of cytokines (ie, IL-2, IL-6, IL-8, IL-10, IL-18, IFN gamma and TNF-alpha). Potential correlations between differential measures of response and the toxicity and efficacy of nivolumab will be explored.
Time Frame: At baseline and at 4 weeks of treatment
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Levels of Peripheral Blood Lymphocyte Phenotype
Description: Humoral and cellular responses to tumor antigens on serum samples will be evaluated by measuring the levels of peripheral blood lymphocyte phenotype. Potential correlations between differential measures of response and the toxicity and efficacy of nivolumab will be explored.
Time Frame: At baseline and at 4 weeks of treatment
Reporting Status: Not Posted

7. Other Pre Specified Outcome: PD-L1 Expression
Description: PD-L1 expression will assist in assessing Overall response rate, PFS, and OS for this treatment.
Time Frame: At baseline and at 4 weeks of treatment
Reporting Status: Not Posted

8. Other Pre Specified Outcome: PD-L2 Expression
Description: PD-L2 expression will assist in assessing Overall response rate, PFS, and OS for this treatment.
Time Frame: At baseline and at 4 weeks of treatment
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Peripheral T Cell Profile Levels
Description: Peripheral T cell profile levels will assist in assessing Overall response rate, PFS, and OS for this treatment.
Time Frame: At baseline and at 4 weeks of treatment
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Serum Interleukin Levels
Description: Serum interleukin levels will assist in assessing Overall response rate, PFS, and OS for this treatment.
Time Frame: At baseline and at 4 weeks of treatment
Reporting Status: Not Posted

11. Post Hoc Outcome: Progression Free Survival Rate at 3 Months and 6 Months
Description: Progression Free Survival (PFS) of nivolumab treatment in patients with metastatic adrenocortical carcinoma is defined as the duration of time from start of treatment to time of documented progression or death, whichever comes first. It will measured per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI scans every 8 weeks. PRS rate at 3 months and 6 months will be calculated as the percentage of patients that have not yet progressed at that timepoint.
Time Frame: At 3 months and 6 months from the initiation of treatment
Measure: Number (95% Confidence Interval); unit: percentage of patients with PFS
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 10
percentage of patients with PFS
  3 Months | 30 [2 to 70]
  6 Months | 20 [0 to 62]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for the study over approximately 1 and a half years with patients being assessed for AEs from the time of treatment initiation, at the beginning of each cycle, through 30 days post last treatment. One cycle equals 28 days and the range of cycles attempted or completed by patients was 1 to 15
Arm/Group | Treatment (Nivolumab)
All-Cause Mortality (participants affected / at risk) | 5/10
Serious Adverse Events (participants affected / at risk) | 7/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Nivolumab) (N=10)
Immune Mediated Hepatitis (Immune system disorders) | 1
Dehydration (Gastrointestinal disorders) | 1 — Patient also with Odynophagia during this event
Sepsis (Infections and infestations) | 1
Vaginal Hemorrhage (Reproductive system and breast disorders) | 1
Progressive Disease/Death (General disorders) | 1 — Patient experienced a thromboembolic event preceding Death
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 — Patient also with fatigue during this SAE
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 — Fatal
Tremor (Nervous system disorders) | 1
Urinary Tract Infection (Infections and infestations) | 1 — Patient also with Confusion during this event
Altered Mental Status (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 — Patient also with Fever during this event
Progressive Disease - Death (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Nivolumab) (N=10)
Anemia (Blood and lymphatic system disorders) | 5
Atrial Flutter (Cardiac disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 2
Adrenal Insufficiency (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Blurred Vision (Eye disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 3
Ascites (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Cheilitis (Gastrointestinal disorders) | 1
Anal Mucositis (Gastrointestinal disorders) | 1
Oral Mucositis (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Odynophagia (Gastrointestinal disorders) | 1
Blisters on lips (Gastrointestinal disorders) | 1
Edema in limbs (General disorders) | 4
Fatigue (General disorders) | 4
Fever (General disorders) | 3
Infusion Related Reaction (General disorders) | 1
Tachypnea (General disorders) | 1
Immune Mediated Hepatitis (Immune system disorders) | 1
Mucosal Infection (Infections and infestations) | 1
Otitis Media (Infections and infestations) | 1
Upper Respiratory Infection (Infections and infestations) | 2
Vaginal Infection (Infections and infestations) | 1
Oral Candidiasis (Infections and infestations) | 1
Alanine Aminotransferase Increased (Investigations) | 2
Alkaline Phosphatase Increased (Investigations) | 3
Aspartate Aminotransferase Increased (Investigations) | 5
Blood Bilirubin Increased (Investigations) | 2
Creatinine Increased (Investigations) | 3
INR Increased (Investigations) | 2
Lymphocyte Count Decreased (Investigations) | 4
Lymphocyte Count Increased (Investigations) | 1
Neutrophil Count Decreased (Investigations) | 1
Weight Loss (Investigations) | 1
White Blood Cell Decreased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 9
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 6
Hypokalemia (Metabolism and nutrition disorders) | 6
Hyponatremia (Metabolism and nutrition disorders) | 5
Back Pain (Musculoskeletal and connective tissue disorders) | 2
Trunk Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1
Right Knee Stiffness (Musculoskeletal and connective tissue disorders) | 1
Hypersomnia (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 1
Chronic Kidney Disease (Renal and urinary disorders) | 1
Urinary Frequency (Renal and urinary disorders) | 1
Gynecomastia (Reproductive system and breast disorders) | 1
Vaginal Hemorrhage (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal Mucositis (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Maculopapular Rash (Skin and subcutaneous tissue disorders) | 3
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 6

LIMITATIONS AND CAVEATS:
The study did not meet its first stage requirements of Interim analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-31): https://cdn.clinicaltrials.gov/large-docs/84/NCT02720484/Prot_SAP_000.pdf